CLINICAL TRIAL: NCT06333678
Title: A Randomized Phase II Study of Sotorasib Versus Continued Consolidation Durvalumab in Patients With KRAS G12C Mutant Locally Advanced Non-small Cell Lung Cancer (LANSCLC) With Persistent ctDNA Defined Minimal Residual Disease
Brief Title: A Study Comparing Sotorasib With Durvalumab in People With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-321
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Sotorasib; Durvalumab; Locally advanced disease; KRAS p.G12C mutation; 22-321
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; sotorasib

STUDY DESIGN:
Intervention Model Description: Phase II randomized trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- continue standard of care (SOC) durvalumab treatment (Active Comparator): Will continue to receive durvalumab, 10 mg/kg IV every 2 weeks or 1500 mg/kg IV every 4 weeks for up to 12 months.
  Interventions: Drug: Durvalumab
- switch sotorasib treatment until progression (Experimental): Will receive sotorasib at 960 mg daily until progression. A dose de-escalation regimen based on toxicity will be implemented as below. If 120 mg cannot be tolerated, sotorasib will be discontinued and the patient will be removed from the trial.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Durvalumab — 10 mg/kg IV every 2 weeks or 1500 mg/kg IV every 4 weeks for up to 12 months.
  Arms: continue standard of care (SOC) durvalumab treatment
Drug: Sotorasib — 960 mg, Patients who do not tolerate sotorasib at 960 mg can be dose reduced to 120 mg.
  Arms: switch sotorasib treatment until progression

SUMMARY:
In this study, the researchers will look at whether having participants switch from durvalumab to sotorasib when they have detectable minimal residual disease (MRD) is an effective treatment approach for locally advanced non-small cell lung cancer (LA-NSCLC). The researchers will see whether this switch to sotorasib can control LANSCLC longer compared to the treatment approach of staying on durvalumab (and not switching to sotorasib).

DETAILED DESCRIPTION:
In the first phase of the randomized trial, defined as the Pre-Monitoring Phase, patients with LANSCLC with a KRAS G12C mutation who are planned to undergo, are undergoing, or very recently completed definitive chemoradiation with the plan for durvalumab consolidation are enrolled. Chemoradiation treatment and all clinical assessments during the Pre-Monitoring Phase are per standard of care as per institutional standards.

Patients who (1) complete chemoradiation, (2) have detectable ctDNA post chemoradiation, (3) are without evidence of progressive disease on imaging, (4) and are planned to start durvalumab consolidation then continue into the Monitoring Phase. All other patients are no longer on trial and are taken off study. Patients in the Monitoring Phase will have ctDNA measured again early-on during durvalumab consolidation (i.e. cycle 3 of durvlalumab +/- 2 weeks) in conjunction with standard of care imaging. Patients with MRD will then continue to the Randomization Phase of trial.

In the Randomization Phase patients will be randomized in a 1:1 fashion to continue standard of care durvalumab (group 1) vs. switch to sotorasib at 960 mg daily (group 2), with the primary endpoint of PFS. Patients switching to sotorasib will undergo a 28-day durvalumab washout and will receive sotorasib at 960 mg daily until progression. Washout will be confirmed by ensuring that cycle 1, day 1 of sotorasib is scheduled for at least 28 days after the most recent durvalumab dose.

ELIGIBILITY:
Inclusion Criteria:

Pre-Monitoring Phase

* Histologic diagnosis of NSCLC
* Locally advanced disease, defined as AJCC 8th Edition Stage III disease.
* Plan for, currently receiving, or recently completed definitive chemoradiation. Definitive radiation is defined as 56-70 Gy in 28-35 fractions concurrently with one of the following chemotherapy regimens:

  * Carboplatin + pemetrexed
  * Cisplatin + pemetrexed
  * Paclitaxel + carboplatin
  * Cisplatin + etoposide
* KRAS p.G12C mutation identified through molecular testing
* Adequate hepatic function, with adequate function defined as AST and ALT < 2.5 x the upper limit of normal (ULN)
* Patient eligible for consolidative durvalumab therapy
* ECOG Performance status 0 - 2.
* Age ≥ 18 years.
* Patients must have decision-making capacity to consent to the study.
* Female subjects must either be of non-reproductive potential (i.e. post-menopausal by history: >/= 55 years old and no menses for 1> year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral salpingectomy OR history of bilateral oophorectomy) or must be willing to comply with contraception requirements.

Monitoring Phase

* Completed definitive chemoradiation. Definitive radiation is defined as 56-70 Gy in 28-35 fractions concurrently with one of the following chemotherapy regimens:

  * Carboplatin + pemetrexed
  * Cisplatin + pemetrexed
  * Paclitaxel + carboplatin
  * Cisplatin + etoposide
* Detectable ctDNA measured within 8 weeks (+2 weeks) of completing definitive chemoradiation
* No evidence of radiographic progression, as measured through SOC imaging, as deemed by principal investigator, including a CT scan of the chest
* ECOG Performance status 0 - 2.
* Plan to start or already started durvalumab consolidation

Therapeutic Phase

* No evidence of radiographic RECIST 1.1 progression, as measured through SOC imaging, as deemed by principal investigator, including a CT scan of the chest
* MRD as measured by ctDNA testing (described above)
* Candidate for sotorasib therapy
* Must have a negative pregnancy test (serum or urine) within 3 days prior to the first dose of sotorasib (if assigned to Group 2).

Exclusion Criteria:

* Serious medical co-morbidities precluding radiotherapy, determined at the discretion of the treating investigator.
* Pregnant or lactating women.
* Physical limitation to undergo radiotherapy.
* Other active malignancy (e.g. receiving active treatment) within the last year except for basal cell carcinoma of the skin and in situ malignancy even if without evidence of disease and patients on adjuvant hormonal therapies (e.g. breast, prostate), or bladder cancer with localized diseases
* Prior pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-01-27 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 3 years
  PFS will be defined as the time from randomization until progression or death , or from the time of randomization until the last follow up imaging (if no progression and alive). Progression will be evaluated by RECIST 1.1 guidelines.

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 1 month after starting Sotorasib
  which we define as a hospitalization, life threatening condition, any death not clearly due to the underlying disease or extraneous causes, or therapy-related grade 3 or higher non-hematologic toxicity. The study will continue if the definition of "acceptable safety" is met.

CONTACTS AND LOCATIONS:
Overall Officials: Narek Shaverdian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - University of Miami (Data Collection Only), Miami, Florida
  - University of Michigan (Data Collection Only), Ann Arbor, Michigan
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York
  - Vanderbilt University (Data Collection Only), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm